CLINICAL TRIAL: NCT06826599
Title: Agreement and Precision Study of UNITY® DX and a Comparator Biometer
Status: Completed | Type: Observational
Sponsor: Cylite Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CYC-CL-SOP-004
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Normal Eyes; Abnormal Eyes
Keywords: Biometric measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Group 1 - Normal Eyes: The eye will be imaged up to seven times with the biometer to achieve three acceptable scans
  Interventions: Device: Investigational Biometer; Device: IOLMaster 700 Biometer
- Group 2 - Eyes with cataracts: The eye will be imaged up to seven times with the biometer to achieve three acceptable scans
  Interventions: Device: Investigational Biometer; Device: IOLMaster 700 Biometer
- Group 3 - Eyes with significant refractive errors: The eye will be imaged up to seven times with the biometer to achieve three acceptable scans
  Interventions: Device: Investigational Biometer; Device: IOLMaster 700 Biometer
- Group 4 - Eyes with abnormal corneal topography: The eye will be imaged up to seven times with the biometer to achieve three acceptable scans
  Interventions: Device: Investigational Biometer; Device: IOLMaster 700 Biometer

INTERVENTIONS:
Device: Investigational Biometer — Investigational non-contact, non-invasive ophthalmic imaging and analysis device used for visualization of ocular structures and measurement of anterior segment and biometric parameters
Device: IOLMaster 700 Biometer — Commercially available non-contact instrument used to capture optical biometry measurements

SUMMARY:
The purpose of this study is to validate the clinical measurement performance of an investigational biometer. Subjects will undergo multiple measurements of the eye, and the agreement, repeatability, and reproducibility of the biometric measurements will be evaluated.

DETAILED DESCRIPTION:
This is intended to be a 1-visit study approximately 3 hours in length with planned duration of exposure of up to 20 minutes per device (investigational biometer and IOLMaster 700). Four cohorts will be enrolled. One eye per subject will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an Institution Review Board approved Informed Consent form.
* Willing and able to attend all scheduled study visits as required by the protocol.
* Identified by the investigator as eligible for at least one of the 4 eye groups identified in the protocol.

Exclusion Criteria:

* Unable to fixate, for example, due to nystagmus or other eye movement abnormality.
* Any ocular disease and/or condition that, in the investigator's clinical judgment, may put the subject at significant risk, may compromise study results, or may interfere significantly with the subject's participation in the study.
* Active ocular infection or inflammation.
* Rigid or contact lens wear during the previous two weeks prior to Screening.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohorts will be selected from approximately one investigative site located in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Central corneal thickness (CCT) | Day 1
  Central corneal thickness will be measured in microns. This outcome measure will be analyzed using Bland-Altman Limits of Agreement, repeatability, reproducibility, and percent coefficient of variation (repeatability and reproducibility) methods.
Lens thickness (LT) | Day 1
  Lens thickness will be measured in microns and analyzed using Bland-Altman Limits of Agreement, repeatability, reproducibility, and percent coefficient of variation (repeatability and reproducibility) methods.
Anterior chamber depth (regression) (ACD-R) | Day 1
  Anterior chamber depth (the physical length from the anterior cornea to the anterior lens) will be measured in microns and analyzed using Bland-Altman Limits of Agreement, repeatability, reproducibility, and percent coefficient of variation (repeatability and reproducibility) methods.
Axial length (regression) (AL-R) | Day 1
  Axial length (the distance between the back and front of the eye) will be measured in millimeters and analyzed using Bland-Altman Limits of Agreement, repeatability, reproducibility, and percent coefficient of variation (repeatability and reproducibility) methods.

SECONDARY OUTCOMES:
Anterior Chamber Depth Sum of Segments (ACD-SoS) | Day 1
  ACD-SoS is calculated by calculating the individual corneal thickness and aqueous depth segments, applying the known refractive indices for each segment, and summing the resultant measurement of each segment. ACD-SoS will be measured in microns and analyzed using Bland-Altman Limits of Agreement, repeatability, and reproducibility methods.
Axial Length Sum of Segments (AL-SoS) | Day 1
  AL-SoS is calculated by calculating the individual corneal thickness, aqueous depth, lens thickness and vitreous length segments, applying the known refractive indices for each segment, and summing the resultant measurement of each segment. AL-SoS will be measured in millimeters and analyzed using using Bland-Altman Limits of Agreement, repeatability, and reproducibility methods.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Ouyang, PhD, Study Director — Cylite Pty Ltd
Locations (1):
- NorthEast Eye Research Associates LLC, Woburn, Massachusetts, United States